CLINICAL TRIAL: NCT04878042
Title: The Negativisation Rate of Positive PCR Swab Tests for the Detection of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) After Treatment With Hydrogen Peroxide: a Double-blind Placebo-controlled Randomised Trial.
Brief Title: COVID-19 Infection Control Using H2O2 Mouth Wash and Nasal Spray
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants
Sponsor: EPISTATA (Network)
Responsible Party: Principal Investigator, Antonio Lazzarino, Director, EPISTATA
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20121617
Record Dates: First submitted 2021-05-04; First posted 2021-05-07 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): Mouth wash and nasal spray containing a diluted solution of hydrogen peroxide
  Interventions: Device: Hydrogen peroxide
- Placebo (Placebo Comparator): Mouth wash and nasal spray not containing a diluted solution of hydrogen peroxide
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Hydrogen peroxide — Mouth wash and nasal spray 3 times a day for 3 days
  Arms: Active
Device: Placebo — Mouth wash and nasal spray 3 times a day for 3 days
  Arms: Placebo

SUMMARY:
Hydrogen peroxide is produced physiologically by oral bacteria and plays a significant role in the balance of oral microecology since it is an important antimicrobial agent. In the epithelial cells, the enzyme superoxide dismutase catalyzes a reaction leading from hydrogen peroxide to the ion superoxide. The induced oxidative stress stimulates a local innate response via activation of the toll-like receptors and the NF-κB. Those kinds of reactions are also activated by viral infections. Virus-induced oxidative stress plays an important role in the regulation of the host immune system and the specific oxidant-sensitive pathway is one of the effective strategies against viral infections. Therefore, nose/mouth/throat washing with hydrogen peroxide may enhance those local innate responses to viral infections. The investigators hypothesised that a treatment with a mouth wash and a nasal spray containing a diluted solution of hydrogen peroxide may accelerate the negativisation rate of a positive PCR swab test for SARS-CoV-2 (COVID-19).

ELIGIBILITY:
Inclusion Criteria:

- recent positive SARS-CoV-2 PCER swab test

Exclusion Criteria:

- severe Covid19 disease

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
The negativisation rate of a positive SARS-CoV-2 (COVID-19) PCR nose swab test | 4 days
  A repeated SARS-CoV-2 PCR nose swab test after a previous positive SARS-CoV-2 PCR nose swab test

CONTACTS AND LOCATIONS:
Overall Officials: Antonio I Lazzarino, MD PhD, Principal Investigator — EPISTATA
Locations (1):
- Clinica Nuova ITOR, Roma, Italy

IPD SHARING:
Plan to Share IPD: No